CLINICAL TRIAL: NCT00976846
Title: Clinical Study Investigating the Performance and Compatibility Characteristics of the Baxter Hollow Fiber Dialyzer Xenium XPH 210 During On-line Hemodiafiltration
Brief Title: Investigation of Performance and Compatibility of the Baxter Dialyzer Xenium XPH 210 During On-line Hemodiafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Praxisverbund Dialyse und Apherese (Other)
Responsible Party: Dr. Peter Ahrenholz, BioArtProducts GmbH, Rostock, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDA-01
Record Dates: First submitted 2009-09-10; First posted 2009-09-15 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: End Stage Kidney Disease
Keywords: hemodialysis; on line; postdilution; high-flux dialyzer; hemodiafiltration
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baxter Xenium XPH 210 (Experimental): Device: Baxter Xenium XPH 210 dialyzer
  Interventions: Device: Dialyzer Baxter Xenium XPH 210

INTERVENTIONS:
Device: Dialyzer Baxter Xenium XPH 210 — High-Flux dialyzer
  Other Names: Baxter Xenium XPH 210

SUMMARY:
The proposed study seeks to determine the appropriate balance between the removal of undesirable small molecular substances (urea, creatinine, phosphate) and large molecular substances (ß2-m) and the retention of important substances (e.g.albumin) for the Baxter Xenium XPH dialyzer type under defined therapeutic conditions of olHDF primarily concerning filtration flow rates in relation to blood flow/plasma water flow rates. Furthermore the possibility of the removal of certain protein-bound substances shall be investigated together with the impact of increasing ultrafiltration on the parameters of the micro-inflammation.

DETAILED DESCRIPTION:
The new high flux dialyser membrane Xenium XPH 210 from Baxter will show an considerably increased removal of ß2-Microglobulin with olHDF in post dilution mode together with a markedly increased removal of small molecules (urea, creatinine, phosphate). The loss of albumin will depend on the treatment modalities. However, the albumin permeability is tolerable over the whole range of total filtration rate selected and applied to the patients.

Together with the albumin loss into the filtrate/dialysate a small amount of albuminbound substances is detectable.

Parameters of micro-inflammation can be influenced by an increasing convective part of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed an informed consent form.
* Patients between 18 and 75 years.
* Patients who have been treated with hemodialysis for more than three months.
* Patients who are treated three times a week for 4-5 hours.
* Patients who are usually treated with high-flux dialyzers.
* Patients who are on a stable anticoagulation and erythropoetin regimen.
* Patients whose hematocrit is over 28 %.
* Patients having no vascular access related problems.

Exclusion Criteria:

* Patients not meeting the inclusion criteria.
* Patients who are in a poor nutritional status as judged by the investigator.
* Patients in a gravid state.
* Patients with an unstable clinical condition (e.g. cardiac or vascular instability).
* Patients whose life expectancy is less than 12 months.
* Patients with a positive anamnesis for the first use syndrome.
* Patients with known coagulation problems.
* Patients who receive hemodialysis via a single dialysis needle or central venous catheter.
* Patients participating in another study that may interfere with the outcome of the present study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Concentration of urea, creatinine, phosphate and ß2-m (pre/post treatment in blood), concentration of albumin (pre/post treatment in blood and dialysate), hematocrit pre/post treatment (for correction of the impact of ultrafiltration on concentrations) | 3 weeks

SECONDARY OUTCOMES:
Pre and post treatment: CMPF (metabolite of furan fatty acids), p-cresol, albumin binding capacity (ABIC) in blood and dialysate, pre and post treatment: IL-6, IL-1ß, sVCAM-1, sICAM-1, CD14+/CD16+, CD62L+, CD11b+ in blood | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Ahrenholz, PhD, Principal Investigator — BioArtProducts GmbH Rostock, Germany
Locations (1):
- Praxisverbund für Dialyse und Apherese, Rostock, Germany